CLINICAL TRIAL: NCT03242278
Title: Real-world Dosing Patterns of Rivaroxaban in the United States (RIVA-D)
Brief Title: Real-world Dosing Patterns of Rivaroxaban in the United States
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18733; XA1511US (Other: Company internal)
Record Dates: First submitted 2017-07-26; First posted 2017-08-08 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation (NVAF); Prevention; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NVAF patients receiving 20 mg rivaroxaban: NVAF patients who receive a standard dose of rivaroxaban (20 mg daily)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- NVAF patients receiving 15 mg rivaroxaban: NVAF patients who receive a reduced dose of rivaroxaban (15 mg daily)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — As prescribed by treating physicians

SUMMARY:
The primary objective is to assess the proportion of Non-valvular atrial fibrillation (NVAF) patients receiving the standard dose of 20 mg of rivaroxaban or the reduced dose of 15 mg of rivaroxaban.

The secondary objective is to determine if dosing patterns for rivaroxaban may be influenced by baseline chronic kidney disease (CKD) status (as a proxy for measured baseline renal function).

ELIGIBILITY:
Inclusion Criteria:

* NVAF (non-valvular atrial fibrillation) will be defined as the occurrence of 2 or more inpatient or outpatient claims with International Classification of Disease ICD-9 427.31 as the diagnosis code at any time in the patient's data history prior to inclusion
* Patients will be required to have 180 days of enrollment for the assessment of baseline characteristics
* CHA2DS2-Vasc score ≥2 during the 180 days prior to index rivaroxaban use baseline period
* Evidence of continuous enrollment in MarketScan during 180 days before the date of the first prescription of rivaroxaban

Exclusion Criteria:

* Patients <18 years of age
* Patients with valvular AF (atrial fibrillation)
* Pregnancy
* Malignant cancers
* Transient cause of AF
* Patients with VTE (Venous thromboembolism), pulmonary embolism or DVT (Deep Vein Thrombosis)
* Patients with major surgery defined as hip or knee replacement
* Prescriptions of OACs (Oral anticoagulants) (apixaban,warfarin, dabigatran, rivaroxaban) before index date
* Prescription of more than one OAC on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation (NVAF)
Sampling Method: Non-Probability Sample
Enrollment: 12507 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Number of NVAF patients receiving 20 mg Rivaroxaban | At baseline
Number of NVAF patients receiving 15 mg Rivaroxaban | At baseline

SECONDARY OUTCOMES:
Baseline renal function | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- New York, New York, United States